CLINICAL TRIAL: NCT04296747
Title: A Single-arm Study Evaluating Efficacy and Safety of Toripalimab Combined With Docetaxel and Cisplatin as Induced Chemotherapy in the Treatment of Localized Hypopharyngeal Squamous Cell Carcinoma
Brief Title: Toripalimab in Combination With Chemotherapy as Induced Chemotherapy for Localized Hypopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO159
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Hypopharyngeal Squamous Cell Carcinoma
Keywords: Toripalimab, hypopharyngeal cancer, induction therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms | interventions — Induction Chemotherapy; Surgical Procedures, Operative; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction therapy (Experimental): patients would accept toripalimab combined with chemotherapy as induction therapy, then radical treatment(surgery or chemoradiotherapy) according to whether the tumor could be resectable or the evaluation result according to RECIST1.1. Ones with PD after induction therapy will enter survival follow-up directly
  Interventions: Drug: induction chemotherapy; Procedure: surgery; Radiation: chemoradiotherapy

INTERVENTIONS:
Drug: induction chemotherapy — Toripalimab 240mg, d1; docetaxel 75mg/m2 d1; cisplatin 75mg/m2 d1, q21d, for 2 cycles
Procedure: surgery — After induction chemotherapy, patients with resectable hypopharyngeal cancer would accept surgery within 2-4 weeks and investigator-selected postoperative treatment
Radiation: chemoradiotherapy — After induction chemotherapy, patients with unresectable hypopharyngeal cancer who achieved CR/PR/SD in the tumor evaluation according to RECIST1.1 would accept another cycle of chemotherapy, and then radical chemoradiotherapy with cisplatin 100mg/m2, q21d

SUMMARY:
60% of hypopharyngeal cancers were locally advanced at the time of diagnosis. The standard treatment was surgery and postoperative radiotherapy. Compared with traditional surgery and postoperative radiotherapy, induction chemotherapy combined with radiotherapy has a better laryngeal retention rate without reducing the curative effect, and established an organ function preservation treatment strategy. Induction chemotherapy can reduce tumor burden and reduce distant metastases. At present, induction chemotherapy followed by concurrent chemoradiotherapy has become the standard treatment for the laryngeal preservation in locally advanced hypopharyngeal and laryngeal cancer. This study aimed to investigate the efficacy and safety of a PD-1 inhibitor toripalimab combined with chemotherapy as induction therapy in hypopharyngeal cancer.

DETAILED DESCRIPTION:
This is a phase II, multicenter, open-label, single-arm study, planned to enroll 100 patients with localized hypopharyngeal squamous cell carcinoma who are newly treated and could accept radical treatment. Patients would be treated with toripalimab combined with docetaxel and cisplatin for two cycles. After the induction chemotherapy is completed, the investigator choose appropriate radical treatment (surgery or chemoradiotherapy) based on tumor evaluation. The primary endpoint is overall objective rate (ORR), the second endpoint include major pathologic response (MPR), 2-year DFS for surgery patients, 2-year PFS for radiotherapy patients, OS and QOL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years when signing informed consent.
2. Pathopharyngeal (histological) confirmed hypopharyngeal squamous cell carcinoma.
3. The initial diagnosis is T1N + M0, T2-4 anyNM0 according to the 8th edition of AJCC.
4. Patients who is suitable and agrees to radical treatment.
5. With evaluable lesions according to the RECIST version 1.1. Note: According to the RECIST 1.1, evaluable lesions refers to a lesion that has been previously treated with radiotherapy. If a clear tumor progression appearance then, it can be used as a measurable lesion.
6. ECOG PS ≤1
7. Adequate organ function, defined as achieving the following laboratory test results ≤ 14 days before treatment

   a. Patients must meet the following laboratory test results: i. ANC ≥ 1.5 x 109 / L ii. Platelets ≥100 x 109 / L iii. Hb ≥90 g / L
   1. Note: Patients must not receive blood transfusion or growth factor within 14 days before blood sample collection due to neutrophil count, platelet, or hemoglobin below study requirements.
   2. Renal function requirements within 4 weeks before treatment: Endogenous creatinine clearance ≥ 60 mL / min or more (based on 24-hour urine creatinine calculation or Cockcroft-Gault formula method).
   3. Serum total bilirubin ≤ 1.5×ULN (Gilbert syndrome patients can be enrolled if the total bilirubin is <3 × ULN).
   4. AST and ALT ≤ 3 × ULN. If the patient has liver metastases, AST and ALT ≤ 5×ULN.
8. Patients with hepatitis B virus (HBV) infection and inactive / asymptomatic HBV carriers; or patients with chronic or active HBV, if HBV DNA <500 IU / mL (or 2500 copies/ mL) will be allowed to enroll. Hepatitis C antibody-positive patients will be allowed to enroll if HCV-RNA is negative during screening.

   NOTE: Patients with detect hepatitis B surface antigen (HBsAg) or HBV DNA, and patients receiving antiviral therapy during screening should be treated for> 2 weeks before enrollment, and Continue treatment for 6 months after study drug therapy
9. Women of childbearing age (WOCBP) must be willing to take effective contraception during the study period and ≥60 days after the last study treatment (including chemotherapy) administration, and the urine or serum pregnancy test result is negative within ≤7 days before treatment.

   a. Women of childbearing age are defined as any woman who has had menarche and has not undergone sterilization (hysterectomy or bilateral ovariectomy) and has not yet reached menopause. Menopause is defined as amenorrhea for 12 months in women> 45 without other biological or physiological causes. In addition, to confirm menopause, women under 55 must have serum follicle stimulating hormone (FSH) levels> 40 mIU / mL.
10. Unsterilized male must be willing to take effective contraception during the study and ≥ 60 days after the last study treatment (including chemotherapy) was administered.

Exclusion Criteria:

1. Not suitable for any of the two-drug chemotherapy prescribed in the protocol
2. Have previously received any treatment for hypopharyngeal squamous cell carcinoma.
3. Patients with evidence of fistula (esophagus / bronchus or esophagus / aorta)
4. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites that require repeated drainage or medical intervention (with clinically significant recurrence requiring additional intervention within 2 weeks after the intervention).
5. Evidence of complete esophageal obstruction that is not suitable for treatment
6. Have been treated with antitumor agents targeted to PD-1, PD-L1 or PD-L2.
7. Have active meningeal disease or uncontrolled brain metastases:

   a. Patients with a history of CNS metastasis while be asymptomatic at the time of screening can be recruit as long as they meet all the following conditions: i. Patients without immediate radiological progression, which means disease progression happened between two consecutive assessments (1 month interval) ii. There are evaluable lesions outside CNS. iii. No need for continuous use of glucocorticoids to treat CNS disease; stable doses of anticonvulsants would be allowed.

   iv. No stereotactic or whole brain radiotherapy was performed within 14 days before treatment.

   b. Patients with new asymptomatic CNS metastases that need to be treated with radiation and / or surgery and have completed corticosteroid therapy.

   i. After treatment, these patients are eligible as long as they meet all other criteria, including those with brain metastases.
8. Patients with active autoimmune disease or history of autoimmune diseases may relapse.

   Note: Patients with the following diseases can be entered for further screening:
   1. Controllable type 1 diabetes
   2. Hypothyroidism (only if it could be controlled by hormone replacement therapy)
   3. Controlled celiac disease
   4. Skin diseases that do not require systemic treatment (eg vitiligo, psoriasis, hair loss)
   5. Any other disease that is not expected to recur without external triggers
9. Any active malignancy within ≤ 2 years before treatment, expect specific cancers which being studied in this study and locally recurrent cancers that have been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical cancer and breast cancer in situ).
10. Any condition requiring systemic treatment with corticosteroids (dose above 10 mg / day of prednisone or equivalent dose of similar agents) or other immunosuppressive agents within ≤ 14 days prior to treatment.

    Note: Patients who are currently or previously using any of the following steroid regimens can be enrolled:
    1. Adrenaline replacement (prednisone ≤10mg / day or equivalent dose of similar agents)
    2. Local, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids with minimal systemic absorption.
    3. Prophylactic short-term (≤7 days) use of corticosteroids (for example, to prevent hypersensitivity caused by contrast agent) or to treat non-autoimmune conditions (for example, delayed-type hypersensitivity reactions caused by exposure to allergens).
11. Have a history of interstitial lung disease, non-infectious pneumonia or uncontrolled disease including pulmonary fibrosis, acute lung disease, etc.
12. Severe chronic or active infections (including tuberculosis infections, etc.) that require systemic antibacterial, antifungal, or antiviral treatment within 14 days of treatment.
13. History of HIV infection.
14. Underwent any major surgery requiring general anesthesia ≤ 28 days before treatment.
15. Previously allogeneic stem cell transplantation or organ transplantation.
16. Have any of the following cardiovascular risk factors:

    1. Cardiogenic chest pain occurs within ≤ 28 days prior to treatment and is defined as moderate pain that limits applianceal activities of daily life.
    2. Symptomatic pulmonary embolism occurred within ≤ 28 days before treatment
    3. Acute myocardial infarction occurred within 6 months before treatment
    4. History of heart failure that has reached New York Heart Association Class III or IV ≤ 6 months before treatment.
    5. Ventricular arrhythmia of grade ≥ 2 occurred within ≤ 6 months before treatment
    6. Cerebrovascular accident occurred within ≤ 6 months before treatment
    7. Uncontrolled hypertension: SBP ≥160 mmHg or DBP ≥100 mmHg, although antihypertensive drugs were used ≤ 28 days before treatment or before the first study drug
    8. Any syncope or convulsions ≤ 28 days before treatment
17. History of severe hypersensitivity to other monoclonal antibodies.
18. Have received Chinese herbal medicine or proprietary Chinese medicine for cancer control within 14 days before the first study drug administration.
19. Live vaccinations within ≤ 4 weeks before treatment. Note: Seasonal flu vaccines are usually inactivated vaccines and are allowed. The vaccine used in the nasal cavity is a live vaccine and is not allowed.
20. Presence of basic medical conditions (including abnormal laboratory test values) or alcohol / drug abuse or dependence that are detrimental to study drug administration or affect drug toxicity or AE interpretation, or that may reduce compliance during the study .
21. Participate in another therapeutic clinical trial at the same time
22. Unintentional weight loss ≥ 5% within 1 month before treatment or severe malnutrition.
23. Nutritional risk index (Shirasu et al 2018) can be used to determine severe malnutrition
24. Pregnant or lactating women
25. peripheral neuropathy ≥ grade 2 at baseline
26. Uncontrolled diabetes, abnormalities of laboratory tests in potassium, sodium or corrected calcium>grade 1 despite standard medication，or hypoalbuminemia ≥ grade 3 within 14 days before treatment.
27. Have received any chemotherapy, immunotherapy (eg interleukin, interferon, thymosin) or any research treatment within 14 days or 5 half-lives (whichever is longer) before the first study drug administration.
28. Other exclusion criteria

    1. Prisoner or jailer.
    2. People who have been compulsorily detained for the treatment of a mental or physical illness, such as an infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
overall objective rate | Up to 2 year
  the percentage of patients whose best overall response was confirmed complete or partial response

SECONDARY OUTCOMES:
major pathologic response | Up to 2 year
  the percentage of patients whose postoperative pathology showing surviving tumor cells ≤10%
2-year overall survival rate | Up to 2 years
  the percentage of patients who survived at 2 year from the first dose
2-year progression-free survival rate | Up to 2 years
  the percentage of patients who accepted chemoradiotherapy and survived without initial radiological progression or death from any cause at 2 year from the first dose
2-year disease-free survival rate | Up to 2 years
  the percentage of patients who accepted surgery and survived without the first appearance of disease or death from any cause at 2 year from the first dose
EORTC H&N 35 form evaluated quality of life | Up to 2 years
  EORTC H&N 35 form evaluated quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Chunmei Bai, Study Chair — Peking Union Medical College Hospital